CLINICAL TRIAL: NCT01807793
Title: Targeted Management Intervention for African-American Men With TIA or Stroke.
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R21NR013001-01A1 (NIH); 1R21NR013001-01A1 (NIH)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Stroke; Transient Ischemic Attack (TIA)
Keywords: Stroke; TIA; African American
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducation (Active Comparator): Psychoeducation will include attending individual and group sessions.
  Interventions: Behavioral: Psychoeducation
- Care as usual (No Intervention): Receive care as usual

INTERVENTIONS:
Behavioral: Psychoeducation
  Arms: Psychoeducation

SUMMARY:
Stroke is the leading cause of disability, third leading cause of death, and one of the most resource-intensive diseases among Americans. African-Americans (AA) have a stroke rate nearly double that of Euro-Americans (EA), and AA who experience a first-ever stroke are younger, have greater stroke disability, more post-stroke complications, and slower recovery compared to EA.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified AA male
* Between 22 and 64 years of age (> age 21 and < age 65).
* Within 6 months of discharge for Stroke /TIA
* Planned or recent home discharge
* Barthel Index (BI) score of > 60
* Available care partner willing to participate
* Be able to speak and understand English

Exclusion Criteria:

* Individuals who are unable or unwilling to provide written informed consent

Ages: 22 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Screening/baseline, 3 months, 6 months
  The primary outcome will be change in medication treatment adherence with stroke risk reduction pharmacotherapies as measured by the Tablets Routines Questionnaire (TRQ)

SECONDARY OUTCOMES:
Biological and health behaviors parameters | Baseline, 3 months, 6 months
  Secondary outcomes are changes in biologic parameters of stroke risk (blood pressure, HbA1c, BMI, cholesterol and triglycerides) and in health behaviors (diet, exercise, smoking, substance use) using standardized instruments

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States